CLINICAL TRIAL: NCT02569697
Title: Development of Adherence Biomarkers for Multiple Microbicide and Multipurpose Prevention Technology (MPT) Dosage Forms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CONRAD (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: D15-135
Record Dates: First submitted 2015-08-21; First posted 2015-10-07 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HEC Placebo Gel (Other): The placebo gel will come in pre-filled individual applicators (4mL). Placebo gel is clear in color and contains HEC as the gel thickener, purified water, sodium chloride, sorbic acid and sodium hydroxide.
  Interventions: Other: HEC Placebo gel
- Placebo Vaginal Insert (Other): The placebo vaginal inserts will be supplied in white plastic bottles. The placebo inserts are white to off-white in color, uncoated and bullet-shaped. The inserts are composed of ingredients generally recognized as safe including isomalt, xylitol, polyvinylpyrrolidone K 30, hydroxypropyl methylcellulose, poloxamer, and sodium stearyl fumarate. The inserts are approximately ½ to 1 inch long and approximately ¼ to ½ inch thick, similar in size to vaginal tablets that are currently available.
  Interventions: Other: Placebo Vaginal Insert
- Placebo Vaginal Film (Other): The placebo vaginal films will be individually wrapped. The placebo vaginal film is a thin, clear to translucent sheet with dimensions of 2 in x 2 in. The ingredients include hydroxyethyl cellulose (HEC), hydroxypropyl methyl cellulose (HPMC, E5), sodium carboxymethyl cellulose (NaCMC), and glycerin.
  Interventions: Other: Placebo Vaginal Film
- Placebo Intravaginal ring (IVR) (Other): The placebo IVRs will be supplied in individual foil pouches. Each ring has a longer white to off-white segment and a shorter transparent/translucent segment, and ingredients include polyurethane, glycerin, water and modified starch.
  Interventions: Other: Placebo Intravaginal Ring

INTERVENTIONS:
Other: HEC Placebo gel
  Arms: HEC Placebo Gel
Other: Placebo Intravaginal Ring
  Arms: Placebo Intravaginal ring (IVR)
Other: Placebo Vaginal Film
  Arms: Placebo Vaginal Film
Other: Placebo Vaginal Insert
  Arms: Placebo Vaginal Insert

SUMMARY:
The purpose of this study is to develop markers for use of placebo vaginal products and measure markers of mucosal semen exposure among healthy women. The study will also monitor safety of placebo product use.

DETAILED DESCRIPTION:
This is a Phase I, non-randomized, open label study in healthy, non-pregnant, HIV negative women, who are not at risk of pregnancy, and are at low risk for STIs (sexually transmitted infections). Participants will be assigned to use one of four placebo products: IVR (intravaginal ring) (approximately 20 participants), and vaginal insert, film or HEC universal placebo gel (approximately 10 participants each). Each woman will provide pre-product use vaginal swabs. Participants assigned to vaginal insert, film or gel will use products with and without timed intercourse with their male partner for a total of two doses of the product, will provide vaginal swabs post product use, and will be seen over 4 visits.

Participants assigned to IVR do not have to be sexually active with a male partner. IVR assigned participants will use a total of 3 IVRs, one at a time. IVR assigned participants will use the first IVR (IVR1) for approximately 24 - 36 hours (no exposure to semen during IVR1 use). IVR assigned participants will use a second IVR (IVR2) for approximately 7 - 10 days and a third IVR (IVR3) for approximately 28 - 32 days. During the use of IVR2 and IVR3, participants may engage in sexual intercourse, but it is not required. Women assigned to IVR use will be seen over 5 visits.

Once a woman completes the study cycle with one study product, she may elect to do another cycle using a different product after a wash-out period of at least 7 days, if she can comply with study product specific protocol requirements. She may elect to do up to four cycles, each with a different study product. For each cycle, V1 screening procedures will be repeated as indicated by symptoms and or participant history, as assessed by the investigator and as outlined in the study manual. If re-screening procedures are not indicated, the new cycle may start with Visit 2 (V2).

At Visit 1 (V1), volunteers will be consented and undergo procedures to confirm they are eligible to continue in the study. Participants will be counseled to refrain from vaginal activity, as applicable, for 48 hours prior to V2.

V2 should occur on days 3 - 10 of the menstrual cycle, or for participants who do not have regular menstrual cycles, when the participant is not having heavy menstrual bleeding. Once it has been confirmed that the participant meets all of the inclusion criteria and none of the exclusion criteria, baseline pre-product use vaginal swabs will be taken. Participants will be required to refrain from any vaginal activity until after Visit 3 (V3).

* Participants assigned to gel, film or insert, will insert one dose (Dose 1) vaginally in the clinic. Vaginal swabs will be obtained in the clinic approximately 15 minutes after product use. Participants will be given vaginal swabs for home use. Participants will be instructed to obtain vaginal swabs, at bedtime daily, for 7 days, starting at the first bedtime after V2. Vaginal swabs will be stored in the participant's refrigerator and returned to the clinic at V3. V3 will occur 7 - 10 days after V2.
* For participants assigned to the IVR, the IVR1 will be inserted by the participant in the clinic. The participant will leave IVR1 in place until V3, which will occur 24 - 36 hours after V2.

At V3:

* Participants assigned to gel, film or insert will return used vaginal swabs to the clinic. Additional vaginal swabs will be obtained in the clinic. Participants will vaginally insert one dose of their assigned product (Dose 2) in the clinic. Vaginal swabs will be obtained in the clinic approximately 15 minutes after product use. The participants will be instructed to have vaginal intercourse with her male sexual partner within approximately 12 hours (± 4 hours) after insertion of the product. They will obtain vaginal swabs, at bedtime daily, for 7 days, starting at the first bedtime after V3 and after timed intercourse, as above. Participants will be instructed to refrain from additional acts of vaginal intercourse or other vaginal activity until Visit 4 (V4). Vaginal swabs will be stored in the participant's refrigerator and returned to the clinic at V4. V4 will occur 7 - 10 days after V3.
* For participants assigned to the IVR, IVR1 will be removed at this visit. Post IVR1 use vaginal swabs will be obtained in the clinic. The second IVR (IVR2) will be inserted by the participant in the clinic. The participant will be instructed to leave the IVR2 in place until V4, which will occur 7 - 10 days after V3. IVR Participants may have vaginal intercourse (not required) during the use of IVR2 but should not have any other vaginal activity during the use of IVR2.

At V4:

* Participants assigned to gel, film or insert will return used vaginal swabs to the clinic. Additional vaginal swabs will be obtained in the clinic. Participants will be exited from the study at this visit or they may elect to use a different study product.
* For participants assigned to the IVR, IVR2 will be removed at this visit. Post IVR2 use vaginal swabs will be obtained in the clinic. The third IVR (IVR3) will be inserted by the participant in the clinic. The participant will leave IVR3 in place until Visit 5 (V5), which will occur 28 - 32 days after V4. Participants may have vaginal intercourse (not required) during the use of IVR3 but should not have any other vaginal activity during the use of IVR3.

At V5 (For IVR only):

• IVR3 will be removed at this visit. Post IVR3 use vaginal swabs will be obtained in the clinic. Participants will be exited from the study at this visit or they may elect to use a different study product.

ELIGIBILITY:
Volunteers must meet all of the following criteria prior to genital sampling at Visit 2:

* Age 18 to 50 years, inclusive
* General good health (by volunteer history and per investigator judgment) without any clinically significant systemic disease (including, but not limited to significant liver disease/hepatitis, gastrointestinal disease, kidney disease, thyroid disease, osteoporosis or bone disease, and diabetes)
* History of Pap smears and follow-up consistent with standard medical practice as outlined in the Study Manual or willing to undergo a Pap smear at V1
* Willing to give voluntary consent and sign an informed consent form
* Willing and able to comply with protocol requirements
* Protected from pregnancy by:

  * hysterectomy
  * reliable methods of contraception other than male or female condoms, contraceptive IVR or male partner's vasectomy
  * abstinence (IVR group only)
  * or in a same sex relationship (IVR group only)
* For gel, insert or film assigned participants: Willing to engage in intercourse with a male sexual partner without the use of male or female condoms as required in the protocol
* For gel, insert or film assigned participants: In a mutually monogamous relationship with a male partner who:

  * Is at least 18 years old
  * Is not known to be HIV positive
  * Has no known risk for STIs
  * Has not undergone a vasectomy
  * Is not known to have azoospermia
  * Is willing and able to comply with protocol requirements regarding sexual activity/ abstinence
  * Can engage with the participant in vaginal intercourse without condoms, as specified in the protocol 8.2. Exclusion Criteria

Volunteers must not meet any of the following criteria prior to genital sampling at Visit 2:

* Currently pregnant
* Currently breastfeeding or planning to breastfeed during the course of the study
* History of sensitivity/allergy to any component of the vaginal products for either the volunteer or her sexual partner, as applicable
* Use of vaginal douches, creams or gels, other than the study product, at any time during the study, beginning 7 days prior to V2
* In the last six months, either the volunteer or her sexual partner (as applicable) diagnosed with or treated for any STI. Note: Women with a history of genital herpes who have been asymptomatic for at least six months may be considered for eligibility
* Positive test for Trichomonas vaginalis, Neisseria gonorrhea, Chlamydia trachomatis or HIV
* Chronic or acute vulvar or vaginal symptoms (pain, irritation, spotting/bleeding, discharge, etc.)
* Known current drug or alcohol abuse which could impact study compliance
* Participation in any other investigational trial within the last 30 days or planned participation in any other investigational trial during the study
* Abnormal finding on laboratory or physical examination or a social or medical condition in either the volunteer or her sexual partner (as applicable) which, in the opinion of the investigator, would make participation in the study unsafe or would complicate interpretation of data

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Presence or absence of spectroscopic pattern signatures or other analytical methods measures of excipient or placebo products or vaginal bacteria in vaginal swabs | 1 - 7 days
Presence or absence of penetration of vaginally-derived biologic analytes or biofilms detected on returned IVRs | 1 - 7 days
Presence or absence of DNA (deoxyribonucleic acid) sequences of SRY (Sex-determining region in the Y chromosome) and TSPY4 (testis-specific protein Y-encoded) | 1 - 7 days
Presence or absence of amelogenin | 1 - 7 days
Changes in dimensions, weight, biologic or chemical composition of IVR | 1 day, 1 week, 1 month
  Assessments in dimensions, weight, biologic or chemical composition will be aggregated to inform changes in overall IVR characteristics

SECONDARY OUTCOMES:
Treatment-emergent adverse experiences among female participants per participant report: urogenital, product related, and/or serious | baseline and at 1 day, 1 week and 1 month
Changes on pelvic exam, as observed by the naked eye | baseline and at 1 day, 1 week and 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Virginia Medical School, Norfolk, Virginia, United States